CLINICAL TRIAL: NCT03576144
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Inhaled Doses of BI 1265162 in Healthy Male Subjects in a Randomised, Double Blind, Placebo-controlled Trial
Brief Title: This Study in Healthy Men Tests How Different Doses of BI 1265162 Are Taken up in the Body and How Well They Are Tolerated.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1399-0002; 2017-001107-71 (EudraCT Number)
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2021-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1265162 (Experimental)
  Interventions: Drug: BI 1265162
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1265162 — Multiple rising inhaled doses
  Arms: BI 1265162
Drug: Placebo — Multiple rising inhaled doses
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1265162 in healthy male subjects following inhalative administration of multiple rising doses.

Secondary objectives is the exploration of the pharmacokinetics (PK) including dose proportionality and time dependency of BI 1265162 after multiple dosing

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Forced expiratory volume in 1 second (FEV1) and Forced vital capacity (FVC) of equal or greater than 80% of predicted normal, at screening and prior to randomisation
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug- Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial- Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* A history of chronic kidney disease (Estimated glomerular filtration rate (EGFR)<59 mls/min including corrections as per ethnicity)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* The subject has a diagnosis history of pulmonary hyperreactivity
* Cannot use Respimat® appropriately
* Male subjects with woman of child bearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 14 days after last administration of trial medication (BI 1265162 or placebo)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Multiple rising dose (MRD) trial was designed as double-blind, randomised, and placebo-controlled within parallel dose groups.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended a specialist site which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Placebo Matching BI 1265162: Participants were administered single and multiple dose of placebo matching BI 1265162 solution for inhalation orally via Respimat® A5 inhaler. On days 1 and 8 participant received a single dose in the morning only. On all other trial days (Days 2 to 7), placebo matching BI 1265162 was administered twice daily.
- 10 Microgram (μg) BI 1265162: Participants were administered single and multiple dose of 10 μg BI 1265162 solution for inhalation orally via Respimat® A5 inhaler. On days 1 and 8 participant received a single dose in the morning only. On all other trial days (Days 2 to 7), 10 μg BI 1265162 was administered twice daily.
- 30 μg BI 1265162: Participants were administered single and multiple dose of 30 μg BI 1265162 solution for inhalation orally via Respimat® A5 inhaler. On days 1 and 8 participant received a single dose in the morning only. On all other trial days (Days 2 to 7), 30 μg BI 1265162 was administered twice daily.
- 100 μg BI 1265162: Participants were administered single and multiple dose of 100 μg BI 1265162 solution for inhalation orally via Respimat® A5 inhaler. On days 1 and 8 participant received a single dose in the morning only. On all other trial days (Days 2 to 7), 100 μg BI 1265162 was administered twice daily.
- 300 μg BI 1265162: Participants were administered single and multiple dose of 300 μg BI 1265162 solution for inhalation orally via Respimat® A5 inhaler. On days 1 and 8 participant received a single dose in the morning only. On all other trial days (Days 2 to 7), 300 μg BI 1265162 was administered twice daily.
- 600 μg BI 1265162: Participants were administered single and multiple dose of 600 μg BI 1265162 solution for inhalation orally via Respimat® A5 inhaler. On days 1 and 8 participant received a single dose in the morning only. On all other trial days (Days 2 to 7), 600 μg BI 1265162 was administered twice daily.
Period: Overall Study
Arm/Group | Placebo Matching BI 1265162 | 10 Microgram (μg) BI 1265162 | 30 μg BI 1265162 | 100 μg BI 1265162 | 300 μg BI 1265162 | 600 μg BI 1265162
Started (Started are treated) | 10 | 8 | 8 | 8 | 8 | 8
Completed | 10 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included included all participants who received at least 1 dose of trial drug. This was the full analysis set population in the sense of International council for harmonisation - efficacy guideline 9: statistical principles for clinical trials (ICH-E9).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 1265162 | 10 Microgram (μg) BI 1265162 | 30 μg BI 1265162 | 100 μg BI 1265162 | 300 μg BI 1265162 | 600 μg BI 1265162 | Total
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.4 (6.9) | 34.0 (4.7) | 27.6 (6.6) | 33.9 (5.6) | 32.4 (6.8) | 35.5 (7.6) | 32.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 8 | 8 | 8 | 8 | 8 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 8 | 8 | 8 | 8 | 8 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 10 | 8 | 8 | 7 | 7 | 8 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events (AEs)
Description: Percentage of participants with drug-related adverse events (AEs).
Time Frame: From first drug administration until 2 days after last drug administration, up to 10 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Placebo Matching BI 1265162 | 10 Microgram (μg) BI 1265162 | 30 μg BI 1265162 | 100 μg BI 1265162 | 300 μg BI 1265162 | 600 μg BI 1265162
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8
Percentage of participants (%) | 0.0 | 12.5 | 12.5 | 50.0 | 50.0 | 12.5

2. Secondary Outcome: Area Under the Concentration-time Curve of the BI 1265162 in Plasma Over the Time Interval of 0 to 12 Hour (h) After Administration of the First Dose (AUC0-12)
Description: Area under the concentration-time curve of the BI 1265162 in plasma over the time interval of 0 to 12 hour (h) after administration of the first dose (AUC0-12).
Time Frame: Pharmacokinetic samples were taken within 1:30 hour:minute (h:m) before dosing and 0:02, 0:05, 0:10, 0:15, 0:20 , 0:40, 1:00, 2:00, 4:00, 8:00 and 12:00 h:m after dosing on day 1.
Population: Pharmacokinetic parameter set (PKS): This subject set included all subjects in the TS who provided at least 1 PK parameter that was not excluded because of protocol deviations relevant to the statistical evaluation of Pharmacokinetic (PK) endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles*Hour Per Litre (pmol*h/L)
Arm/Group | 10 Microgram (μg) BI 1265162 | 30 μg BI 1265162 | 100 μg BI 1265162 | 300 μg BI 1265162 | 600 μg BI 1265162
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Picomoles*Hour Per Litre (pmol*h/L) | 82.5 (24.5) | 226 (23.2) | 734 (22.5) | 2430 (35.2) | 6320 (21.3)
Statistical Analysis 1: Comparison: 10 Microgram (μg) BI 1265162 vs 30 μg BI 1265162 vs 100 μg BI 1265162 vs 300 μg BI 1265162 vs 600 μg BI 1265162; Dose proportionality for AUC0-12 of BI 1265162 in plasma was assessed using a power model (regression model applied to log-transformed data). The corresponding ANCOVA model included the logarithm of the dose as a covariate. No statistical hypotheses were tested in a confirmatory sense; Test type: Other; ANCOVA; Slope = 1.0474, 90% CI 2-sided [0.9997 to 1.0951], Standard Error of Mean 0.0283 — Standard Error of the mean is actually standard error of slope.Based on the estimate for the slope parameter (β), a 2-sided 90% CI for the slope was computed. Perfect dose proportionality would correspond to a slope of 1

3. Secondary Outcome: Maximum Measured Concentration of the BI 1265162 in Plasma After Administration of the First Dose (Cmax)
Description: Maximum measured concentration of the BI 1265162 in plasma after administration of the first dose (Cmax).
Time Frame: Pharmacokinetic samples were taken within 1:30 hour: minute (h:m) before dosing and 0:02, 0:05, 0:10, 0:15, 0:20, 0:40, 1:00, 2:00, 4:00, 8:00, 12:00 and 24:00 h:m after dosing on day 1.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles Per Litre (pmol/L)
Arm/Group | 10 Microgram (μg) BI 1265162 | 30 μg BI 1265162 | 100 μg BI 1265162 | 300 μg BI 1265162 | 600 μg BI 1265162
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Picomoles Per Litre (pmol/L) | 55.2 (36.1) | 158 (27.4) | 391 (24.4) | 1330 (43.5) | 4000 (28.0)
Statistical Analysis 1: Comparison: 10 Microgram (μg) BI 1265162 vs 30 μg BI 1265162 vs 100 μg BI 1265162 vs 300 μg BI 1265162 vs 600 μg BI 1265162; Dose proportionality for Cmax of BI 1265162 in plasma was assessed using a power model (regression model applied to log-transformed data). The corresponding ANCOVA model included the logarithm of the dose as a covariate. No statistical hypotheses were tested in a confirmatory sense; Test type: Other; ANCOVA; Slope = 1.0091, 90% CI 2-sided [0.9451 to 1.0732], Standard Error of Mean 0.0380 — Standard Error of the is actually standard error of slope. Based on the estimate for the slope parameter (β), a 2-sided 90% CI for the slope was computed. Perfect dose proportionality would correspond to a slope of 1

4. Secondary Outcome: Area Under the Concentration-time Curve of the BI 1265162 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of the BI 1265162 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss).
Time Frame: Pharmacokinetic samples were taken 0:05 hour: minute (h:m) before dosing and 0:02, 0:05, 0:10, 0:15, 0:20, 0:40, 1:00, 2:00, 4:00, 8:00 and 12:00 h:m after last dosing on day 8.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles*Hour Per Litre (pmol*h/L)
Arm/Group | 10 Microgram (μg) BI 1265162 | 30 μg BI 1265162 | 100 μg BI 1265162 | 300 μg BI 1265162 | 600 μg BI 1265162
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Picomoles*Hour Per Litre (pmol*h/L) | 104 (18.8) | 284 (40.0) | 1190 (29.4) | 3800 (29.3) | 7010 (36.4)
Statistical Analysis 1: Comparison: 10 Microgram (μg) BI 1265162 vs 30 μg BI 1265162 vs 100 μg BI 1265162 vs 300 μg BI 1265162 vs 600 μg BI 1265162; Dose proportionality for AUCτ,ss of BI 1265162 in plasma was assessed using a power model (regression model applied to log-transformed data). The corresponding ANCOVA model included the logarithm of the dose as a covariate. No statistical hypotheses were tested in a confirmatory sense; Test type: Other; ANCOVA; Slope = 1.0520, 90% CI 2-sided [0.9972 to 1.1069], Standard Error of Mean 0.0325 — Standard Error of the mean is actually standard error of slope. Based on the estimate for the slope parameter (β), a 2-sided 90% CI for the slope was computed. Perfect dose proportionality would correspond to a slope of 1

5. Secondary Outcome: Maximum Measured Concentration of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss).
Time Frame: as for outcome 4
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles Per Litre (pmol/L)
Arm/Group | 10 Microgram (μg) BI 1265162 | 30 μg BI 1265162 | 100 μg BI 1265162 | 300 μg BI 1265162 | 600 μg BI 1265162
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Picomoles Per Litre (pmol/L) | 55.6 (25.7) | 143 (38.5) | 640 (42.7) | 1710 (35.5) | 3670 (39.9)
Statistical Analysis 1: Comparison: 10 Microgram (μg) BI 1265162 vs 30 μg BI 1265162 vs 100 μg BI 1265162 vs 300 μg BI 1265162 vs 600 μg BI 1265162; Dose proportionality for Cmax,ss of BI 1265162 in plasma was assessed using a power model (regression model applied to log-transformed data). The corresponding ANCOVA model included the logarithm of the dose as a covariate. No statistical hypotheses were tested in a confirmatory sense; Test type: Other; ANCOVA; Slope = 1.0361, 90% CI 2-sided [0.9722 to 1.1001], Standard Error of Mean 0.0379 — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 2 days after last drug administration, up to 10 days.
Arm/Group | Placebo Matching BI 1265162 | 10 Microgram (μg) BI 1265162 | 30 μg BI 1265162 | 100 μg BI 1265162 | 300 μg BI 1265162 | 600 μg BI 1265162
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/10 | 1/8 | 2/8 | 5/8 | 4/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 1265162 (N=10) | 10 Microgram (μg) BI 1265162 (N=8) | 30 μg BI 1265162 (N=8) | 100 μg BI 1265162 (N=8) | 300 μg BI 1265162 (N=8) | 600 μg BI 1265162 (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT03576144/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03576144/SAP_001.pdf